CLINICAL TRIAL: NCT06685211
Title: A Randomized, Sham Controlled, Masked Study to Evaluate the Efficacy of Alternating Current Stimulation Using the Eyetronic System for the Treatment of Glaucoma
Brief Title: Electrical Stimulation for Vision Neuroenhancement in Glaucoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: EYETRONIC, Inc (Unknown)
Responsible Party: Principal Investigator, Jeffrey L Goldberg, Professor and Chair of Ophthalmology, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 76900
Record Dates: First submitted 2024-11-09; First posted 2024-11-12 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Glaucoma; Glaucoma Open-Angle
Keywords: glaucoma; open-angle glaucoma
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- rtACS treatment (Experimental): Participants will receive 10 days of rtACS treatment in office.
  Interventions: Device: Eyetronic rtACS
- Sham (Placebo Comparator): Participants will be wearing device but no stimulation will occur for 10 treatments in office.
  Interventions: Device: Sham rtACS

INTERVENTIONS:
Device: Eyetronic rtACS — The repetitive, transorbital alternating current stimulation (rtACS) is a device for non-invasive Interventional Neurophysiology. The electrical charge and current density applied during rtACS safe and able to modulate existing neuronal elements in the eye and brain.
  Arms: rtACS treatment
Device: Sham rtACS — Participants will wear the Eyetronic system but there will be no active stimulations applied.
  Arms: Sham

SUMMARY:
The purpose of the study is to evaluate the efficacy, transorbital alternating current stimulation (rtACS) using the EYETRONIC for the treatment in patients with glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be at least 18.
* Participant must has the ability to comply with the requirements of the study and complete the schedule of events (SOE).
* Participant's clinical diagnosis must be consistent with primary open angle glaucoma (including but not limited to normal tension, low tension or general open angle) characterized by the following features: Mean deviation (MD) worse than -6 but better than -20 on reliable Humphrey Visual Field 24-2 testing
* Participant's eye pressure must be clinically stable, with IOP < 18.
* If a participant has two eyes meeting study criteria, the worse eye as determined by visual field index (VFI) or patient preference, will be deemed includable. If both eyes qualify and have the same VFI, the patient may choose which eye they are willing to enter, or else a randomization procedure will assign one eye to the study.
* Participant must understand and sign the informed consent. If the participant's vision is impaired to the point where he/she cannot read the informed consent document, the document will be read to the participant in its entirety.

Exclusion Criteria:

* Participant is unable to comply with study procedures or follow-up visits.
* Participant has a history of ocular herpes zoster.
* Participant has a requirement of acyclovir and/or related products during study duration. To be eligible for this study, the participant must discontinue use of these products prior to enrollment and must not continue with the products until after they have completed the study.
* Participant has evidence of corneal opacification or lack of optical clarity.
* Participant has uveitis or other ocular inflammatory disease.
* Participant is receiving systemic steroids or other immunosuppressive medications.
* Participant is currently participating in or has within the last 3 months participated in any other clinical trial of a drug by ocular (if in the study eye) or systemic administration.
* Participant is pregnant or lactating.
* Participant has, in the opinion of the investigator, any physical or mental condition that would increase the risk of participation in the study or may interfere with the study procedures, evaluations and outcome assessments.
* Patients with opened skull, after trepanation or with heart and brain pacemaker.
* Patients with implanted intracranial metals such as clippings, coilings, ventriculo-peritoneal shunts, endoprosthesis etc.
* Patients with any skin damage in the area of electrode placement.
* Children and comatose patients.
* Patients with recent history of epileptic seizure.
* Patients with uncontrolled high levels of blood pressure (<160 mmHg) or uncontrolled high levels of intraocular pressure (<27 mmHg).
* Patients abusing drugs or alcohol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Field Index (VFI) | 3 Months
  Measuring the change in the Visual Field Index (VFI) from baseline to month 3.
Mean Deviation (MD) | 3 Months
  Measuring the change in Mean Deviation on Visual Field from Baseline to Month 3.
Pointwise Linear Regression (PLR) | 3 Months
  Measuring the PLR of the visual field points from baseline to Month 3.

SECONDARY OUTCOMES:
Ganglion Cell Layer | 3 Months
  The change in ganglion cell layer as measured by optical coherence tomography (OCT) through 3 months
Retinal Nerve Fiber Layer | 3 Months
  The change in nerve fiber layer thickness as measured by OCT through 3 months
Best Corrected Visual Acuity | 3 Months
  The change in best corrected visual acuity (BCVA) through 3 months
Stead-State Visually Evoked Potential | 3 Months
  The change in visual evoked potential (VEP) through 3 months
OCT-Angiography | 3 Months
  The change in OCT angiography (OCT-A) through 3 months
Retinal Metabolic Analysis | 3 Months
  The change in retinal metabolic analysis (RMA)/OcuMet imaging through 3 months
Visual Field indicies in Non-Study Eye | 3 Months
  Change in visual field indices in non-study eye through 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Goldberg, MD PhD, Principal Investigator — Stanford University
Locations (1):
- Byers Eye Institute at Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR